CLINICAL TRIAL: NCT06577649
Title: From Pain in the Face to Perceptual Distortion: Exploring Mechanisms and Novel Treatment Strategies
Brief Title: Pain and Perceptual Distortion of Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5771
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Neuropathic Pain; Orofacial Pain
Keywords: Repetitive transcranial magnetic stimulation; N-of-1 trials; Perceptual distortion; Post-traumatic trigeminal neuropathic pain
MeSH Terms: conditions — Neuralgia; Facial Pain

STUDY DESIGN:
Intervention Model Description: "n-of-1" single-blinded randomized controlled cross-over design: (A) active-sham-active-sham or (B) sham-active-sham-active.
Who Masked: Participant
Masking Description: The order of interventions (A) active-sham-active-sham or (B) sham-active-sham-active were randomized using a computer-based random sequence generation program. The allocation was conducted by a nurse not involved in the project and consisted of 12 sealed, opaque and numbered envelopes consisting of information about the treatment order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): Continuous theta burst stimulation
  Interventions: Device: Active repetitive transcranial magnetic stimulation (rTMS)
- Sham group (Sham Comparator): Sham repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (sham rTMS)

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation (rTMS) — cTBS (50 Hz, 600 pulses, 80% resting motor threshold) for 40s was applied continuously as active rTMS at the face representation area of primary somatosensory cortex (S1)
  Arms: Active group
Device: Sham repetitive transcranial magnetic stimulation (sham rTMS) — A sham rTMS was applied using the same stimulation parameters as with cTBS, but using a placebo coil, which produced similar sound as the real coil.
  Arms: Sham group

SUMMARY:
Post-traumatic trigeminal neuropathic pain (PTNP) is "a unilateral or bilateral facial or oral pain following and caused by trauma to the trigeminal nerve(s), with other symptoms and/or clinical signs of trigeminal nerve dysfunction, and persisting or recurring for more than 3 months". PTNP may result from a major craniofacial/oral trauma or may be subsequent to relatively minor dental treatments such as teeth extractions, surgeries, root canal treatment. Patients suffering from this condition have a significantly reduced quality of life. Unfortunately, the currently available management modalities are associated with limited success and side effects.

Repetitive transcranial magnetic stimulation (rTMS), which is a safe, non-invasive brain stimulation technique has emerged as a potential treatment for chronic pain. In this study, the purpose is to explore the potential of rTMS in treating the persistent neuropathic pain by providing individualized treatment for the sufferers.

DETAILED DESCRIPTION:
In addition to pain, a curious observation in people with PTNP is that they report that the painful facial area is "swollen" or "feels differently". There are often no clinical signs or physical differences present, hence such self-reported "illusions" may represent a kind of disrupted body image or a "perceptual distortion" of the face and can be speculated to contribute to the maintenance of facial pain. rTMS paradigms are being widely applied in both therapeutic and investigative studies.In this project, the aim is to employ continuous theta-burst stimulation (cTBS), an inhibitory rTMS paradigm, to evaluate its effect on pain perception and PD in people with PTNP.

In this project, people with PTNP (N=9) received a rTMS (50 Hz, 600 pulses for 40s) session/week as intervention for four consecutive weeks at the primary somatosensory cortex (face area) in a "n-of-1" single-blinded randomized controlled cross-over design: (A) active-sham-active-sham or (B) sham-active-sham-active. That is the same participant received both active and sham either in the (A) order or (B). Pain intensity and perceptual distortion (PD) as perceived size changes of the affected face area were measured at baseline, immediately, 60 mins after rTMS in each session and end of the session (a week after rTMS), one and three months after rTMS. Questionnaires on quality of life, jaw function, sleep quality were also assessed. Changes in pain and PD after each intervention were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Persistent Post-traumatic trigeminal neuropathic pain patients for 6 months or longer
* Stable on analgesic medication

Exclusion Criteria:

* past history of TMS therapy or TMS-related contraindications (pacemaker, epilepsy etc.).
* Major stroke
* Pregnancy
* Severe organic brain damage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention).
  Changes in pain intensity from baseline to end of each session measured using self-reported pain dairy using a 0-10 visual analog scale (VAS; 0=no pain and 10=worst pain imaginable). The intervention (active and sham rTMS) were each given in 2 sessions. In total, the participant received 4 sessions of intervention.
Changes in perceptual distortion | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention).
  Perceptual distortion defined as perceived change in the size/shape of the affected face area will be measured using Numerical Rating Scale ranging from -100% through 0% to +100%, where 0% = no size change, -100% = half the size and +100% = double the size in comparison with non-affected side of face and drawings of the affected area. The changes will be measured from baseline to the end of each session as done for pain intensity.

SECONDARY OUTCOMES:
Changes in sleep quality | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Measured using the Pittsburgh Sleep Quality Index (PSQI-DK). Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Changes in perceived health or health related quality of life | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Will be measured using Short Form Survey-36- (SF -36).The instrument includes scales for physical functioning, social functioning, role limitations due to physical or emotional problems, mental health, energy, pain and general health perception. It consists of 36 items. Each item is graded on a scale of 0 to 100, with 0 and 100 serving as the lowest and highest possible scores respectively. A high score corresponds to better health status.
Changes in oral-health related quality of life | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Will be measured using Oral Health Impact Profile (OHIP-14) questionnaire .The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse and lower scores indicate better oral health related quality of life (OHRQol).
Changes in functional limitation of the jaw. | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Will be measured using jaw functional limitation scale (JFLS-20). The scores range from 1 to 200, with higher scores indicating deteriorating jaw function.
Changes in Psychological Distress | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Will be measured using general anxiety disorder (GAD-7) scale. Total score is obtained by adding score for each question (total points). A score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder.
Changes in Pain Catastrophizing | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Will be measured using the Pain Catastrophizing Scale (PCS-DK). Consists of 13 items. Each item is ranged from 0-4. A high score corresponds to a high degree of pain catastrophizing.
Changes in patients health | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Measured using patient health questionnaire-15 (PHQ-15).Each item on the PHQ-15 is rated on a 3-point scale (0=not bothered at all; 1=bothered a little; 2= bothered a. lot). The total score can range from 0 to 30, with higher scores indicating greater severity of somatic symptoms.
Changes in neuropathic pain characteristics | Prior to intervention at each session (baseline) to the end of that session (7 days after intervention), 1 and 3 months after intervention.
  Measured using modified PainDetect questionnaire. The PainDetect questionnaire was slightly modified so that the oral components can also be added. It is scored from 0 to 38, with total scores of less than 12 considered to represent nociceptive pain, 13-18 possible neuropathic pain, and >19 representing >90% likelihood of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Simple F Kothari, BDS, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Department of Dentistry and Oral Health, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kothari SF, Dagsdottir LK, Kothari M, Blicher JU, Kumar A, Buchholtz PE, Ashkanian M, Svensson P. Effect of repetitive transcranial magnetic stimulation on altered perception of One's own face. Brain Stimul. 2020 May-Jun;13(3):554-561. doi: 10.1016/j.brs.2020.01.001. Epub 2020 Jan 8. PMID 32289676